CLINICAL TRIAL: NCT05460572
Title: Cardiac Metabolic Profiling in the Fed State
Acronym: CAMP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University Medical Center Groningen (Other)
Collaborators: Netherlands Heart Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 202100291
Record Dates: First submitted 2022-07-05; First posted 2022-07-15 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Heart Failure
Keywords: Cardiac Metabolism; Arteriovenous gradient; Metabolites; Fed State; Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients undergoing PVI procedure and who are treated with peripheral parental nutrition (Other): Patients undergoing elective PVI procedure who will receive peripheral parental nutrition before start of the procedure.
  Interventions: Dietary Supplement: Peripheral Parental Nutrition

INTERVENTIONS:
Dietary Supplement: Peripheral Parental Nutrition — Peripheral parenteral nutrition (PPN) through an intravenous (iv) line

SUMMARY:
This is a non-randomized interventional prospective study, aiming to provide insight into cardiac substrate utilization in the fed state. Patients will participate during an elective PVI procedure which would have taken place regardless of the current study. During this study, study subjects will receive peripheral parenteral nutrition (PPN) through an intravenous (iv) line. During the procedure, blood samples will be drawn from the catheters which will be in situ for the purpose of the elective PVI procedure. Cardiac arteriovenous (A-V) gradients of metabolites will be measured, reflecting cardiac uptake and release of metabolites in the fed state.

DETAILED DESCRIPTION:
The heart requires tremendous amounts of energy to sustain its continuous mechanical work. The heart can utilize various metabolic substrates to generate energy, including carbohydrates, lipids, amino acids and ketone bodies. However, most research on cardiac fuel use has been done in rodents and surprisingly little is known about cardiac fuel use in patients with heart disease. Prior experimental studies showed that carbohydrates are important fuels for cardiac energy production. In contrast, a recent study in patients with heart disease showed that the heart only utilizes little amounts of carbohydrates. This study was however, performed in fasting subjects, which could have an important effect on substrate preference. The primary aim of this non-randomized interventional prospective study is to provide insight into cardiac substrate utilization in the fed state. Patients will participate during an elective PVI procedure which would have taken place regardless of the current study. During this study they will receive peripheral parenteral nutrition (PPN) through an intravenous (iv) line. Blood samples will be drawn with the catheters which will already be in situ for the purpose of the elective PVI procedure. Cardiac arteriovenous (A-V) gradients of metabolites will be measured, reflecting cardiac uptake and release of metabolites in the fed state.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing elective PVI procedure
* Adult age (≥ 18 years)
* Have given verbal and written informed consent

Exclusion Criteria:

* Chronic renal disease with an estimated glomerular filtration rate (eGFR) <30 mL/min/1.73 m2
* Chronic liver disease and/or severe liver dysfunction with ASAT and/or ALAT > 3x the upper limit of normal (ULN)
* Pregnancy or breastfeeding
* Insulin dependent diabetics
* Congenital metabolic disease
* Weight below 40 kg
* Inability to understand and read Dutch or English
* Known allergy or hypersensitivity to any of the non-investigational products in the study protocol
* Any other clinical condition that would jeopardize patient's safety while participating in this trial or may prevent the patient from adhering to the trial protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-07-15 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Quantitative analysis of cardiac uptake and release of metabolites in the fed state | Peripheral Parental Nutrition will start before start of the PVI procedure. Sixty minutes after start of peripheral parental nutrition, blood sampling will be performed.
  Cardiac fuel use will be mapped by metabolomics on blood from the left atrium, the coronary sinus and the right atrium during PVI procedure. By comparing the concentrations of metabolites in the blood from different anatomical locations, cardiac uptake or release of energy substrates will be determined.

SECONDARY OUTCOMES:
Quantitative analysis of uptake and release of metabolites in the fed state in the lower extremity | Peripheral Parental Nutrition will start before start of the PVI procedure. Sixty minutes after start of peripheral parental nutrition, blood sampling will be performed.
  Fuel use will be mapped by metabolomics on blood from the left atrium and the femoral vein during PVI procedure. By comparing the concentrations of metabolites in the blood from different anatomical locations, the uptake or release of metabolites by the lower extremity will be determined.
  Comparisons will be made between arterial blood (left atrium) and venous blood from the leg (femoral vein), in order to quantify extraction or secretion of each metabolite.
Differences in cardiac uptake and release of metabolites between heart failure patients with reduced, mid-range and preserved ejection fraction and patients without HF | Peripheral Parental Nutrition will start before start of the PVI procedure. Sixty minutes after start of peripheral parental nutrition, blood sampling will be performed.
  Cardiac fuel use will be mapped by metabolomics on blood from the left atrium, the coronary sinus and the right atrium during PVI procedure. By comparing the concentrations of metabolites in the blood from different anatomical locations, cardiac uptake or release of energy substrates will be determined. To determine differences in arteriovenous gradients between HF with reduced, mid-range and preserved ejection fraction versus patients without HF, patients will be assigned to one of the following four groups based on available information about presence of heart disease and most recently documented ejection fraction in the EPD.

CONTACTS AND LOCATIONS:
Overall Officials: Daan Westenbrink, MD PhD, Principal Investigator — Universitary Medical Center Groningen
Locations (1):
- Universitary Medical Center Groningen, Groningen, Netherlands